CLINICAL TRIAL: NCT02302404
Title: A Single-centre, Randomized, Double-blind (Sponsor Unblinded), Placebo-controlled Two-part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK2982772, in Single (in Both Fed and Fasted States) and Repeat Oral Doses in Healthy Male Subjects
Brief Title: A Safety and Tolerability Study of GSK2982772, in Single (in Both Fed and Fasted States) and Repeat Oral Doses in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Clinical Unit at Cambridge (Addenbrooks) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200975
Record Dates: First submitted 2014-10-27; First posted 2014-11-27 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Inflammatory Bowel Diseases
Keywords: FTIH; pharmacodynamics; pharmacokinetics; GSK2982772; safety; Repeat dose; tolerability
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — GSK2982772

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1: GSK2982772 Single Ascending Dose (Part A) (0.1-10mg) (Experimental): Eight subjects will be randomized equally (1:1:1:1) to one of the 4 placebo-controlled dose sequences with 2 subjects in each sequence and each subject having four dose periods (3 active dose of GSK2982772 + 1 placebo dose). The subjects will fast overnight from Day -1 to Day 1 of the treatment period. Two of the 8 subjects will be randomized to the dosing on Day 1 as sentinel dosing. Assuming adequate safety in the judgment of the Principal Investigator (e.g., vital signs, ECGs, and adverse events) through approximately 24 hours; the remaining 6 subjects may be randomized to dosing on the following day. Subjects will receive single planned doses of GSK2982772 as 0.1, 0.5, 2.5, and 10mg. A sequential design will be used including approximately weekly dose escalations while allowing for a sufficient washout period. The proposed doses may be adjusted based on emerging safety and PK
  Interventions: Drug: GSK2982772 solution; Drug: GSK2982772 capsule; Drug: Placebo solution; Drug: Placebo capsule
- Cohort 2: GSK2982772 Single Ascending Dose (Part A) (40-240mg) (Experimental): Eight subjects will be randomized equally to one of the 4 placebo-controlled dose sequences with 2 subjects in each sequence and each subject having 4 dose periods (3 active dose of GSK2982772 +1 placebo dose). The subjects will fast overnight from Day -1 to Day 1 of the treatment period. Two of the 8 subjects will be randomized to the dosing on Day 1 as sentinel dosing. Assuming adequate safety in the judgment of the Principal Investigator (e.g., vital signs, ECGs, and adverse events) through 24 hours; the remaining 6 subjects may be randomized to dosing on the following day. Subjects will receive single planned doses of GSK2982772 as 40, 100, 180, and 240 mg. A sequential design with weekly dose escalations and sufficient washout period will be used. The proposed doses may be adjusted based on emerging safety and PK. After the completion of the fasted treatment periods, subjects will receive a high fat meal within 30 minutes of dosing with GSK2982772 during a final treatment period.
  Interventions: Drug: GSK2982772 capsule; Drug: Placebo capsule
- Cohort 3: GSK2982772 Repeat Dose (Part B) (Experimental): Twelve subjects will be randomized to repeat doses of GSK2982772 or placebo in a 3:1 ratio. The subjects will fast overnight from Day -1 to Day 1 and overnight from Day 13 to Day 14. The selection of appropriate daily doses will be performed upon consideration of available safety and tolerability and PK data from Part A. Once-daily dosing is planned, but twice-daily dosing may be considered based upon the exposure observed in the Part A data
  Interventions: Drug: GSK2982772 capsule; Drug: Placebo capsule
- Cohort 4: GSK2982772 Repeat Dose (Part B) (Experimental): Twelve subjects will be randomized to repeat doses of GSK2982772 or placebo in a 3:1 ratio. The subjects will fast overnight from Day -1 to Day 1 and overnight from Day 13 to Day 14. The selection of appropriate daily doses will be performed upon consideration of available safety and tolerability and PK data from Part A and/or any preceding repeat dose cohorts in Part B. Once-daily dosing is planned, but twice-daily dosing may be considered based upon the exposure observed in Part A or any preceding repeat dose cohorts in Part B
  Interventions: Drug: GSK2982772 capsule; Drug: Placebo capsule
- Cohort 5: GSK2982772 Repeat Dose (Part B) (Experimental): Twelve subjects will be randomized to repeat doses of GSK2982772 or placebo in a 3:1 ratio. The subjects will fast overnight from Day -1 to Day 1 and overnight from Day 13 to Day 14. The selection of appropriate daily doses will be performed upon consideration of available safety and tolerability and PK data from Part A and/or any preceding repeat dose cohorts in Part B. Once-daily dosing is planned, but twice-daily dosing may be considered based upon the exposure observed in the Part A or any preceding repeat dose cohorts in Part B.
  Interventions: Drug: GSK2982772 capsule; Drug: Placebo capsule
- Cohort 6: GSK2982772 Single Ascending Dose (Part A) (Experimental): This additional cohort in Part A of the study will only be conducted to allow for evaluation of additional dose levels or repeated evaluation of a dose level already studied. Doses will be selected based on the safety, tolerability, and PK data from Part A and/or previous Part B cohorts. Eight subjects will be randomized equally (1:1:1:1) to one of the 4 placebo-controlled dose sequences with 2 subjects in each sequence and each subject having four dose periods (3 active dose of GSK2982772 + 1 placebo dose). The selection of appropriate daily doses will be performed upon consideration of available safety and tolerability and PK data from Part A and/or any preceding repeat dose cohorts in Part B.
  Interventions: Drug: GSK2982772 capsule; Drug: Placebo capsule
- Cohort 7: GSK2982772 Repeat Dose (Part B) (Experimental): This additional cohort in Part B of the study will only be conducted to allow for evaluation of additional dose levels or repeated evaluation of a dose level already studied Doses will be selected based on the safety, tolerability, and PK data from Part A and/or previous Part B cohorts. Twelve subjects will be randomized to repeat doses of GSK2982772 or placebo in a 3:1 ratio. The selection of appropriate daily doses will be performed upon consideration of available safety and tolerability and PK data from Part A and/or any preceding repeat dose cohorts in Part B.
  Interventions: Drug: GSK2982772 capsule; Drug: Placebo capsule

INTERVENTIONS:
Drug: GSK2982772 solution — Clear, colorless solution containing GSK2982772 in water with 5% ethanol (0.1mg/mL). Administered orally in required volumes for dosing less than 5mg
  Arms: Cohort 1: GSK2982772 Single Ascending Dose (Part A) (0.1-10mg)
Drug: GSK2982772 capsule — Size 00 White Opaque capsule containing GSK2982772 as white to almost white solid. Administered orally with water for dosing from 5 to 120 mg
Drug: Placebo solution — Clear, colorless solution containing placebo in water with 5% ethanol (0.1mg/mL). Administered orally in required volumes for dosing less than 5mg
  Arms: Cohort 1: GSK2982772 Single Ascending Dose (Part A) (0.1-10mg)
Drug: Placebo capsule — Size 00 White Opaque capsule containing Placebo as white to almost white solid

SUMMARY:
This study is the first administration of GSK2982772 in humans. The study will evaluate the safety, tolerability, pharmacokinetics (PK), and exploratory pharmacodynamics (PD) of single and repeat oral doses of up to 14 days with GSK2982772 in healthy male subjects.

This study is planned to include approximately 52 subjects and will consist of 2 parts: Part A - single ascending dose, randomized, placebo controlled, 4 way crossover. In addition to the crossover treatment periods, up to 8 subjects in cohort 2 will participate in an additional treatment period and receive GSK2982772 with a high-fat meal. Part B - repeat dose, randomized, placebo controlled, sequential-group. In both cohorts of Part A (Cohorts 1 and 2), subjects will be randomized equally (1:1:1:1) to one of 4 treatment sequences. Within each period, allocation of active to placebo treatment will be 3:1.

In all cohorts in Part B (Cohorts 3, 4 and 5) subjects will be randomized to GSK2982772 or placebo in a 3:1 ratio. If required, subjects in the additional cohorts in Part A (Cohort 6) and Part B (Cohort 7) will be randomized to GSK2982772 or placebo in a 1:1:1:1 and 3:1 ratio, respectively. The study duration, including screening and follow-up, is not expected to exceed 105 days for any subject in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, neurological examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Note: Screened subjects with laboratory values outside of the normal range may be repeated once for inclusion into the study at the discretion of the Investigator.
* Body weight >= 50 kilogram (kg) and body mass index (BMI) within the range 19 - 30 (kilogram/squared meter) kg/m^2 (inclusive).
* Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until at least five half-lives of study medication after the last dose of study medication or the follow-up visit, whichever is longer. a. Abstinence, defined as sexual inactivity consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception; b. Vasectomy with documentation of azoospermia; c. Male condom plus partner use of one of the contraceptive options: Contraceptive subdermal implant that meets the standard operation procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Oral Contraceptive, either combined or progestogen alone. Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches; Occlusive cap (female diaphragm or cervical/vault cap) with a vaginal spermicide (foam, gel, cream or suppository). These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The Investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and as explained by the investigator.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of active infections within 14 days of receiving study medication.
* Average QT duration corrected for heart rate by Fridericia's formula (QTcF) > 450 milliseconds (msec) of three measures taken at least 5 minutes apart in the semi-supine position.
* History or diagnosis of obstructive sleep apnoea.
* History of a significant respiratory disorder.
* History or current evidence of febrile seizures, epilepsy, convulsions, significant head injury, or other significant neurologic conditions.
* Unable to refrain from prescription or non-prescription drugs, including agents active in the central nervous system, vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and throughout the study, unless in the opinion of the Investigator and/or GlaxoSmithKline Medical Monitor (if needed) the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study, defined as: For United Kingdom (UK) - an average weekly intake of >21 units for males. One unit is equivalent to 8 gram(g) of alcohol: a half-pint (approximately 240 millilitre [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Current use or history of regular tobacco- or nicotine-containing product use within 6 months of screening. Subject must have urinary cotinine levels indicative of non-smoking status at screening visit.
* Unwilling or unable to swallow multiple size 00 capsules as part of study participation
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator and/or Medical Monitor (if appropriate), contraindicates their participation.
* Subject received a vaccine (either live attenuated or non-live) within 30 days of randomization OR plan to receive a live attenuated vaccine within 30 days + 5 half-lives of the last dose of study medication.
* Subjects with impaired renal function defined as Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine > 1.6 milligram/decilitre (mg/dL) with an age appropriate glomerular filtration rate (GFR) <=60 (millilitre/minute [mL/min]/1.73 squared meter [m^2]) estimated by the CKD-EPI equation.
* A positive anti-nuclear antibody (ANA) or elevated C-reactive protein (CRP) outside of the normal reference range.
* Peripheral capillary oxygen saturation (SpO2) < 95% at room air.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. As potential for and magnitude of immunosuppression with this compound is unknown, subjects with presence of hepatitis B core antibody (HBcAb) should also be excluded.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* A positive tuberculosis test.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Part B Specific Exclusion Criteria:

* Total cholesterol >=300 mg/dL or triglycerides >=250 mg/dL. - Subjects who, in the Investigator/designee's judgment, pose a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behavior and/or any evidence of suicidal ideation on any questionnaires (e.g., type 4 or 5 on the Columbia Suicide Severity Rating Scale [C-SSRS] in the last 5 years).
* For Cohort 5 Only (or another Cohort where Entero Test is to be performed) - History of gall bladder surgery or gall bladder removal, or history of an acute disease state (e.g., cholelithiasis) within 14 days of receiving study medication.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2016-03-05 (Actual); Study Completion 2016-03-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSK2982772 as assessed by clinical monitoring and reporting of adverse events (AE) and serious adverse events (SAE) | Up to approximately 105 days
  AEs and SAEs will be collected from the start of Study Treatment until the follow-up contact
Change in laboratory values after single (fed and fasted) and repeat doses of GSK2982772 | Up to approximately 105 days
  Laboratory assessments will include analysis of hematology parameters, clinical chemistry, routine urinalysis, lipid panel (Part B Only) and other screening Tests
Electrocardiogram (ECG) assessment after single (fed and fasted) and repeat doses of GSK2982772 | Up to approximately 105 days
  12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals. Triplicate 12-lead ECGs will be obtained pre-dose on Day 1 and Day 14 (Part B only).
Change in vital signs after single (fed and fasted) and repeat doses of GSK2982772 | Up to approximately 105 days
  Vital signs will be measured in semi-supine position after short period of time (e.g., 5 to 10 minutes rest) and will include systolic and diastolic blood pressure, temperature, pulse rate, pulse oximetry (SpO2), and respiratory rate. Triplicate vital signs will be obtained pre-dose on Day 1 and Day 14 (Part B only)
Summary of physical examinations after single (fed and fasted) and repeat doses of GSK2982772 | Up to approximately 105 days
  A complete physical examination will include assessment of the Cardiovascular, Respiratory, Gastrointestinal and Neurological systems. Weight will also be measured and recorded. A brief physical examination will include assessments of the skin, lungs, cardiovascular system, abdomen (liver and spleen), and assessment for lymphadenopathy

SECONDARY OUTCOMES:
Composite of derived Pharmacokinetic (PK) parameters of GSK2982772 measured by AUC (0-t), AUC (0-infinity), Cmax, Tmax and t1/2,following single (fed and fasted) doses | Pre-dose, Days 1 (20 and 40 minutes, 1, 1.5, 2, 3, 5, 8, 10 and 12 hours), 2 and 3 post dose
  PK parameters for GSK2982772 will include area under the blood drug concentration versus time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC [0-t]), area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC [0-infinity]), maximum observed blood drug concentration (Cmax), time to maximum observed blood drug concentration (Tmax), and terminal half-life (t1/2) following single (fed and fasted) doses, where data allow
Composite of derived blood PK parameters of GSK2982772 measured by AUC (0-t), AUC (0-infinity), AUC (0-tau), Cmax, Tmax and t1/2,following repeat doses | Pre-dose, Days 1 (20 and 40 minutes, 1, 1.5, 2, 3, 5, 8, 10 and 12 hours) , 2, 3, 4, 5, 6, 7, 14 (20 and 40 minutes, 1, 1.5, 2, 3, 5, 8, 10 and 12 hours), 15 and 16 post-dose
  Derived blood PK parameters for GSK2982772 will include AUC(0-t), AUC(0-infinity), area under the concentration-time curve over the dosing interval (AUC [0-tau]), Cmax, Tmax and t1/2, following single and repeat doses
Estimation of accumulation ratio (Ro) of GSK2982772 following single and repeat doses | Up to Day 14 of Part B
  Ro will be calculated as the ratio of AUC(0-24) (Repeat Dose) to AUC(0-24) (Single Dose). Day 14 (Repeat Dose) will be compared with Day 1 (Single Dose) in order to estimate the accumulation ratio for each dose level
Ratio of Plasma 4beta-hydroxycholesterol to cholesterol during pre-treatment and following repeat dosing of GSK2982772 | Up to Day 14 of Part B
  A comparison will be made between the ratio of 4beta-hydroxycholesterol: cholesterol at baseline and on Day 14 to assess potential changes in cytochrome P450 isoform 3A4(CYP3A4) enzyme activity following GSK2982772 treatment.
Ex-vivo GSK2982772 blood:plasma concentration ratio over a range of concentrations and % blood cell association. | Up to approximately 105 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- [Derived] Weisel K, Scott NE, Tompson DJ, Votta BJ, Madhavan S, Povey K, Wolstenholme A, Simeoni M, Rudo T, Richards-Peterson L, Sahota T, Wang JG, Lich J, Finger J, Verticelli A, Reilly M, Gough PJ, Harris PA, Bertin J, Wang ML. Randomized clinical study of safety, pharmacokinetics, and pharmacodynamics of RIPK1 inhibitor GSK2982772 in healthy volunteers. Pharmacol Res Perspect. 2017 Dec;5(6):e00365. doi: 10.1002/prp2.365. PMID 29226626
- See also: Results for study 200975 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/200975?search=study&b'search_terms=200975'#rs